CLINICAL TRIAL: NCT00539695
Title: Phase II Trial Using Low Dose IL-2 to Induce Regulatory T Cells in Patients After Allogeneic Hematopoietic Stem Cell Transplantation as Graft Versus Host Disease Prophylaxis
Brief Title: Low Dose IL-2, Hematopoietic Stem Cell Transplantation, IL2 for GVHD
Acronym: IL2 for GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rayne Rouce, Assistant Professor of Pediatrics, Hem-Onc Cell & Gene, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-20971-IL2 for GvHD; IL-2 for GVHD (Other: Baylor College of Medicine)
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Acute Lymphoblastic Leukemia; ALL; Acute Myelogenous Leukemia; AML; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Myeloproliferative Disorder; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Non-malignant Diseases Requiring Allogeneic HSCT
Keywords: Stem Cell transplant; Graft verus host disease; IL-2; acute lymphoblastic leukemia; ALL; acute myelogenous leukemia; AML; chronic myelogenous leukemia; myelodysplastic syndrome; myeloproliferative disorder; Hodgkin lymphoma; non-Hodgkin lymphoma; non-malignant diseases requiring allogeneic HSCT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Myeloproliferative Disorders; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IL2 Administration (Experimental): SCHEDULE OF IL-2 ADMINISTRATION: Patients will receive a fixed dose (1x10e5 units/m2/dose) of IL-2 given as a subcutaneous injection three times weekly (separated by at least one day) for 6 weeks beginning no earlier than day +7 after HSCT but beginning no later than 30 days after HSCT.
  Time will be measured as 'week beginning with first IL-2 injection.'
  T cell Induction via IL-2 to reduce GVHD
  Interventions: Biological: IL-2

INTERVENTIONS:
Biological: IL-2 — IL2 Administration:
  Patients will be given a fixed dose (1x10e5 units/m2/dose) of IL-2 given as a subcutaneous injection three times weekly (separated by at least one day) for 6 weeks beginning no earlier than day +7 after HSCT but beginning no later than 30 days after HSCT. If the patient has not developed >grade I side effects to IL-2 and has not developed >grade I GVHD then the patient may continue the IL-2 for 6 additional weeks. Time will be measured as 'week beginning with first IL-2 injection.
  Other Names: Proleukin; Aldesleukin; Interleukin-2

SUMMARY:
Patients are being asked to participate in this study because treatment for their disease requires a stem cell transplant (SCT). Stem cells are the source of normal blood cells found in the bone marrow and lead to recovery of blood counts after bone marrow transplantation. With stem cell transplants, regardless of whether the donor is a full match to the patient or not, there is a risk of developing graft-versus-host disease (GVHD).

GVHD is a serious and sometimes fatal side effect of SCT. GVHD occurs when the new donor stem cells (graft) recognizes that the body tissues of the patient (host) are different from those of the donor. When this happens, cells in the graft may attack the host organs. How much this happens and how severe the GVHD is depends on many things, including how different the donors cells are, the strength of the drugs given in preparation for the transplant, the quality of transplanted cells and the age of the person receiving the transplant.

Typically, acute GVHD occurs in the first 100 days following transplant, while chronic GVHD occurs after day 100. Acute GVHD most often involves the skin, where it can cause anywhere from a mild rash to complete removal of skin; liver, where it can anywhere from a rise in liver function tests to liver failure; and the gut, where it can cause anywhere from mild diarrhea to profuse, life-threatening diarrhea. Most patients who develop GVHD experience a mild to moderate form, but some patients develop the severe, life-threatening form.

Previous studies have shown that patients who receive SCT's can have a lower number of special T cells in their blood, called regulatory T cells, than people who have not received stem cell transplants. When regulatory T cells are low, there appears to be an increased rate of severe, acute GVHD. A drug known as IL-2 (Proleukin) has been shown to increase the number of regulatory T cells in patients following stem cell transplant, and in this study investigators plan to give low dose IL-2 after transplant.

This study is called a phase II study because its major purpose is to find out whether using a low-dose of IL-2 will be effective in preventing acute GVHD. Other important purposes are to find out if this treatment helps the patient's immune system recover regulatory T cells faster after the transplant. This study will assess the safety and toxicity of low-dose IL-2 given to patients after transplantation and determine whether this drug is helpful in preventing GVHD.

DETAILED DESCRIPTION:
Participation in this protocol will last about 1 year.

To participate in this study, the patient will need to have undergone a stem cell transplant. Before the treatment starts, investigators would like to test the patient's blood blood for the number of regulatory T cells already present before beginning IL-2.

Treatment Plan:

Before the conditioning treatment for the transplant, 30 to 40 ml (6 to 8 teaspoonfuls) of blood will be collected from the patient for regulatory T cell analysis. Approximately same amount of blood will also be collected on day 0 (the day of the transplant), and at the following times after the transplant: day 7 (the day the IL-2 will most likely start) then weekly for another eleven weeks, then monthly for 8 months.

On approximately day 7 following the transplant, if the patient is well and meets the eligibility requirements, the IL-2 injections will begin. These will be given subcutaneously (as a small injection just under the skin) three times per week for 6 weeks. The injections may also been given through a special catheter, called an Insuflon catheter, that is placed just under the skin for a week at a time. The first dose must be given in the hospital, but the remaining doses can be given at home. The patient will be taught how to give the injections to him/ herself.

If the patient's body has no serious toxicities from the IL-2 and has not developed severe GVHD, the patient can continue to get the injections the same way for an additional 6 weeks. If at any time the patient develops severe GVHD or serious toxicity related to the IL-2,the injections will be stopped. If the patient's disease returns (relapse) or he or she does not engraft (accept the donor graft), the patient will be removed from the study.

The patient's labs will be followed closely while he/she is receiving the IL-2 injections, as well as heart, kidney and lung functions; however, these are all standard tests that the patient will receive after transplant regardless of participation in this study.

ELIGIBILITY:
INCLUSION CRITERIA:

INCLUSION CRITERIA FOR INITIAL STUDY ENROLLMENT:

Patients will be eligible for initial enrollment on this study as long as they meet the following criteria:

* Diagnosis of acute lymphoblastic leukemia, acute myelogenous leukemia, chronic myelogenous leukemia, myelodysplastic syndrome, myeloproliferative disorder, Hodgkin lymphoma, non-Hodgkin lymphoma or non-malignant disease requiring allogeneic HSCT
* Birth to age 70 years of age
* Study entry consent is signed and faxed to Research Coordinator

INCLUSION CRITERIA AT TIME OF IL-2 ADMINISTRATION:

* At least day +7 post transplant
* Less than or equal to 30 days post transplant
* Lansky or Karnofsky score greater than or equal to 50%
* Total bilirubin less than or equal to 1.5mg/dL
* Alanine aminotransferase level (ALT) less than or equal to five times normal, serum direct bilirubin less than or equal to 1.5mg/dL, albumin greater than or equal to 3.0gm/dL
* Serum creatinine less than three times normal or creatinine clearance greater than 80mg/min/1.73m2
* Ensure that informed consent signed and faxed to Research Coordinator

EXCLUSION CRITERIA:

EXCLUSION CRITERIA AT TIME OF IL-2 ADMINISTRATION:

Patients will be ineligible to receive IL-2 injections if any of the following is true:

* Active, acute GVHD greater than or equal to grade II
* Serious, active bacterial, fungal or viral infection (i.e. intensive care)
* Clinical Signs of severe pulmonary dysfunction
* Clinical Signs of sever cardiac dysfunction
* Receiving corticosteroids as GVHD treatment
* Hypersensitivity or allergy to IL-2

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rayne Rouce, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Kennedy-Nasser AA, Ku S, Castillo-Caro P, Hazrat Y, Wu MF, Liu H, Melenhorst J, Barrett AJ, Ito S, Foster A, Savoldo B, Yvon E, Carrum G, Ramos CA, Krance RA, Leung K, Heslop HE, Brenner MK, Bollard CM. Ultra low-dose IL-2 for GVHD prophylaxis after allogeneic hematopoietic stem cell transplantation mediates expansion of regulatory T cells without diminishing antiviral and antileukemic activity. Clin Cancer Res. 2014 Apr 15;20(8):2215-25. doi: 10.1158/1078-0432.CCR-13-3205. Epub 2014 Feb 26. PMID 24573552

RESULTS

PARTICIPANT FLOW:
Groups:
- IL2 Administration: SCHEDULE OF IL-2 ADMINISTRATION: Patients will receive a fixed dose (1x10e5 units/m2/dose) of IL-2 given as a subcutaneous injection three times weekly (separated by at least one day) for 6 weeks beginning no earlier than day +7 after HSCT but beginning no later than 30 days after HSCT.
  Time will be measured as 'week beginning with first IL-2 injection.'
  T cell Induction via IL-2 to reduce GVHD
  IL-2: IL2 Administration:
  Patients will be given a fixed dose (1x10e5 units/m2/dose) of IL-2 given as a subcutaneous injection three times weekly (separated by at least one day) for 6 weeks beginning no earlier than day +7 after HSCT but beginning no later than 30 days after HSCT. If the patient has not developed >grade I side effects to IL-2 and has not developed >grade I GVHD then the patient may continue the IL-2 for 6 additional weeks. Time will be measured as 'week beginning with first IL-2 injection.
Period: Overall Study
Arm/Group | IL2 Administration
Started | 25
Evaluable Patients | 22 (Patients who received IL-2.)
Completed | 12
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | IL2 Administration
Number analyzed (Participants) | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  less than 20 yrs | 13 [9 to 15]
  greater and equal 20 yrs | 47.5 [30.5 to 59.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicities
Description: Assessment of the safety and the toxicity of low-dose IL-2, administered according to the dosage described in this protocol, in this group of patients The outcome measure is the proportion of participants with dose limiting toxicities.
Time Frame: 6-12 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants of DLT
Arm/Group | IL2 Administration
Number analyzed (Participants) | 22
proportion of participants of DLT | 0.045 [0.001 to 0.228]

2. Secondary Outcome: Rate of Severe (Grade III or IV) Acute GVHD
Description: To determine the efficacy of low-dose IL-2 in the prevention of severe (grade III or IV) acute GVHD
Time Frame: Up to 12 weeks on low-dose IL-2
Population: Participants received low-dose IL-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IL2 Administration
Number analyzed (Participants) | 22
percentage of participants | 4.5 [0.12 to 22.8]

3. Secondary Outcome: Percentage Change in CD4+ CD25+ FoxP3+ Regulatory T Cells (Tregs) From Pre to Post IL-2 Infusions
Description: To investigate the immunomodulatory effects of IL-2 administered after allogeneic hematopoietic stem cell transplantation
Time Frame: 12 weeks
Population: Participants received low-dose IL-2 and had pre and post IL-2 Treg measurements.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | IL2 Administration
Number analyzed (Participants) | 16
percentage | 55.6 [-37.8 to 417.7]

4. Other Pre Specified Outcome: Ancillary Studies
Description: To conduct ancillary studies on those patients to investigate before, during and after IL-2 administration to determine:
  * The immunophenotype of PBMCs
  * The suppressive activity of CD4+ CD25+ FoxP3+ Tregs
  * Cytokines secreted by PBMCs
  * NK cell analysis
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IL2 Administration
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL2 Administration (N=22)
Anorexia (Gastrointestinal disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1) — constitutional symptoms
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) — Constitutional Symptoms
Gastrointestinal - Other: Gall Bladder (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1)
Infection - Other: GNR Line Infection (B Cepacia complex) (Infections and infestations) | 1 (1)
Infection - Other: Gastrointestinal_Abdomen (Infections and infestations) | 1 (1)
Infection - Other: Parainfluenza (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL2 Administration (N=22)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 9 (48)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 13 (48)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 12 (42)
Alkaline phosphatase (Metabolism and nutrition disorders) | 3 (8)
Anorexia (Gastrointestinal disorders) | 2 (3)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 5 (16)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (11)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 14 (67)
Constipation (Gastrointestinal disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (12)
Creatinine (Metabolism and nutrition disorders) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 11 (31)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (11)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Edema: head and neck (Blood and lymphatic system disorders) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 3 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (13)
Fatigue (lethargy, malaise, asthenia) (Gastrointestinal disorders) | 8 (14)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 9 (31)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 7 (27)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (11)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Cardiac disorders) | 3 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 2 (4)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 3 (3)
Insomnia (General disorders) | 2 (2)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (5)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9 (30)
Mood alteration - Anxiety (Nervous system disorders) | 2 (4)
Mood alteration - Depression (Nervous system disorders) | 2 (3)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2 (5)
Nausea (Gastrointestinal disorders) | 18 (50)
Neuropathy: sensory (Nervous system disorders) | 5 (7)
PTT (Partial Thromboplastin Time) (General disorders) | 3 (4)
Pain - Abdomen NOS (General disorders) | 8 (11)
Pain - Back (General disorders) | 3 (3)
Pain - Bone (General disorders) | 3 (4)
Pain - Head/headache (General disorders) | 10 (18)
Pain - Joint (General disorders) | 2 (2)
Pain - Other: Abdomen (General disorders) | 2 (5)
Pain - Other: Dysuria (General disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (9)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (6)
Pulmonary/Upper Respiratory - Other: Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13 (27)
Renal/Genitourinary - Other: Dysuria (Renal and urinary disorders) | 2 (2)
Rigors/chills (General disorders) | 3 (4)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 (24)
Tremor (Nervous system disorders) | 2 (2)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 12 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes